CLINICAL TRIAL: NCT06387667
Title: Unveiling the Fungal Frontier: Characterizing Diversity and Antifungal Resistance in Immunocompromised ICU Patients With Respiratory Tract Infections
Brief Title: Characterizing Diversity and Antifungal Resistance in Immunocompromised ICU Patients With Respiratory Tract Infections
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New Valley University (Other)
Responsible Party: Principal Investigator, Asmaa Nady Hussein, Lecturer of Internal Medicine, New Valley University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FIRTI
Record Dates: First submitted 2024-04-01; First posted 2024-04-29 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Immunocompromised ICU Patients With Respiratory Tract Infections
MeSH Terms: interventions — Blood Cell Count; Microscopy; Sensitivity and Specificity

STUDY DESIGN:
Intervention Model Description: Immunocompromised ICU Patients with Respiratory tract infections
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immunocompromised ICU patients (Experimental): Immunocompromised ICU Patients with Respiratory tract infections
  Interventions: Diagnostic Test: Complete blood count; Diagnostic Test: C-reactive protein, urea, creatinine, Random blood glucose (RBG), aspartate aminotransferase (AST), alanine aminotransferase (ALT); Radiation: CT chest; Diagnostic Test: Microscopic examination; Diagnostic Test: culture and sensitivity

INTERVENTIONS:
Diagnostic Test: Complete blood count — blood sample
Diagnostic Test: C-reactive protein, urea, creatinine, Random blood glucose (RBG), aspartate aminotransferase (AST), alanine aminotransferase (ALT) — serum sample
Radiation: CT chest — Computed tomography of the chest
Diagnostic Test: Microscopic examination — sputum and bronchoalveolar lavage (BAL)
Diagnostic Test: culture and sensitivity — for bacterial and fungal

SUMMARY:
Immunocompromised individuals face a heightened risk of life-threatening fungal infections, which arise from a multitude of environmental and commensal fungi. Surveillance data from ICUs worldwide identifies Candida spp. as the dominant foe, responsible for 80% of such infections, earning it the dubious distinction of being the third most prevalent pathogen. While C. albicans holds the dubious crown as the most common Candida offender, recent years have witnessed a concerning trend toward non-Albicans candida, raising concerns about potential antifungal resistance.

DETAILED DESCRIPTION:
For critically ill patients in the ICU, the threat of invasive fungal infections is a hidden danger, particularly in the presence of any of the following opportunistic factors:

(A) Pre-existing lung disease: Idiopathic pulmonary fibrosis (IPF) , Chronic obstructive pulmonary disease (COPD), or Sarcoidosis.

(B) Patient comorbidities:

1. Immunosuppression: Neutropenia, Corticosteroid therapy, Immunosuppressive medication for inflammatory or autoimmune diseases; T-cell suppressants: Antithymocyte globulin (ATG), Calcineurin inhibitors (e.g., tacrolimus, cyclosporine) or B-cell suppressants: Rituximab, Severe sepsis (immune paralysis): Inherited severe immunodeficiency: Chronic granulomatous disease (CGD), Wiskott-Aldrich syndrome (WAS), and Common variable immunodeficiency (CVID) or Acquired immunodeficiency due to HIV/AIDS.
2. Underlying medical conditions: Liver failure, Diabetes mellitus, or cardiovascular disease.
3. Viral Pneumonia: Influenza-associated pulmonary aspergillosis (IAPA) and Coronavirus disease 2019 (COVID-19)
4. Hematological and solid malignancies.
5. Hematopoietic stem cell transplantation (HSCT).
6. Prior fungal exposure: Aspergillus colonization before or during ICU admission .

(C) Environmental factors: Construction work, Geo-climatic factors, Tobacco or cannabis use, Air, food, or spice contamination, Gardening activity or occupation.

For diagnosing an invasive fungal infection (IFI), symptoms are unspecific; fever, cough, or chest pain and often missed in patients on corticosteroids, the host criteria including the presence of high-risk factors like neutropenia, malignancies, or immunosuppression, the clinical criteria; specific imaging findings on chest X-ray, high-resolution computed tomography (HRCT) or bronchoscopy indicating pulmonary involvement then finally mycological Criteria: Positive fungal detection in samples (culture, polymerase chain reaction 'PCR', GM).

In Non-Hematological Patients, diagnosis often delayed due to atypical symptoms and imaging, potentially leading to airway invasion vs. angioinvasion, differing clinical presentation and tests. Also, Lower GM yield compared to hematological patients. Crucially, this delayed diagnosis contributes to the higher mortality in non-hematological patients. This underscores the urgent need to establish improved diagnostic capabilities for invasive pulmonary aspergillosis using mycological tests in non-hematological individuals.

By closely monitoring the prevalence and drug susceptibility patterns of fungal pathogens, leads to acquiring crucial insights into their dynamics and refine the therapeutic approaches accordingly. This data empowers clinicians to make informed decisions regarding antifungal therapy, minimizing unnecessary drug exposure and preserving the effectiveness of the antifungal weapons.

Based on the need for more specific studies on diagnosis, prophylaxis, and therapy of critically ill, non-neutropenic, patients, and the significant threats of fungal infections to immunocompromised patients, particularly in ICU settings, understanding the diversity and antifungal resistance of these infections is crucial for optimizing treatment strategies and improving patient outcomes. This study will provide valuable insights into the epidemiology and antifungal resistance of fungal infections in immunocompromised ICU patients, informing the development of more effective prevention and treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (aged >18 years old) admitted to the Assiut University Hospital's intensive care units with pneumonia and hospitalized patients who developed hospital-acquired or ventilator-associated pneumonia who don't respond to antibiotics for 48 hours or with a CT finding suspected for fungal pneumonia.

Patients included must have at least one of the following conditions as a contributor to immunocompromise:

* Pre-existing lung disease: IPF, COPD, or sarcoidosis.
* Immunosuppression: Neutropenia, on corticosteroids, or immunosuppressive drugs, inherited or acquired immunodeficiency.
* Underlying comorbidities: (Diabetes Mellitus,Chronic kidney disease, Liver cirrhosis)
* Malignancy (Hematological or solid)

Exclusion Criteria:

* Patients refused to contribute to the study.
* Unsatisfactory sample.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of fungal species causing pneumonia in immunocompromised ICU patients | baseline

SECONDARY OUTCOMES:
Determine the antifungal susceptibility profiles of the identified fungal isolates. | baseline
Number of associated specific patient factors with the type or antifungal resistance of fungal infections | baseline

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sprute R, Nacov JA, Neofytos D, Oliverio M, Prattes J, Reinhold I, Cornely OA, Stemler J. Antifungal prophylaxis and pre-emptive therapy: When and how? Mol Aspects Med. 2023 Aug;92:101190. doi: 10.1016/j.mam.2023.101190. Epub 2023 May 17. PMID 37207579
- [Background] Kett DH, Azoulay E, Echeverria PM, Vincent JL; Extended Prevalence of Infection in ICU Study (EPIC II) Group of Investigators. Candida bloodstream infections in intensive care units: analysis of the extended prevalence of infection in intensive care unit study. Crit Care Med. 2011 Apr;39(4):665-70. doi: 10.1097/CCM.0b013e318206c1ca. PMID 21169817
- [Background] Bassetti M, Garnacho-Montero J, Calandra T, Kullberg B, Dimopoulos G, Azoulay E, Chakrabarti A, Kett D, Leon C, Ostrosky-Zeichner L, Sanguinetti M, Timsit JF, Richardson MD, Shorr A, Cornely OA. Intensive care medicine research agenda on invasive fungal infection in critically ill patients. Intensive Care Med. 2017 Sep;43(9):1225-1238. doi: 10.1007/s00134-017-4731-2. Epub 2017 Mar 2. PMID 28255613
- [Background] Meersseman W, Lagrou K, Maertens J, Van Wijngaerden E. Invasive aspergillosis in the intensive care unit. Clin Infect Dis. 2007 Jul 15;45(2):205-16. doi: 10.1086/518852. Epub 2007 Jun 13. PMID 17578780
- [Background] Hage CA, Carmona EM, Evans SE, Limper AH, Ruminjo J, Thomson CC. Summary for Clinicians: Microbiological Laboratory Testing in the Diagnosis of Fungal Infections in Pulmonary and Critical Care Practice. Ann Am Thorac Soc. 2019 Dec;16(12):1473-1477. doi: 10.1513/AnnalsATS.201908-582CME. No abstract available. PMID 31526275